CLINICAL TRIAL: NCT00967772
Title: A Clinical Trial to Investigate the Safety/Tolerability and Pharmacokinetics of Naftopidil After Oral Administration in Korean Healthy Male Volunteers
Brief Title: The Safety/Tolerability and Pharmacokinetics (PKs) of Naftopidil in Korean Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FLV100
Record Dates: First submitted 2009-08-26; First posted 2009-08-28 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Safety; tolerability
MeSH Terms: interventions — naftopidil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Naftopidil (Experimental)
  Interventions: Drug: Naftopidil

INTERVENTIONS:
Drug: Naftopidil — 25mg/ 50 mg/ 75mg dosage tablets

SUMMARY:
The safety/tolerability and pharmacokinetics (PK) of Naftopidil (commercial name: Flivas) after oral administration will be investigated in Korean healthy male volunteers. All volunteers will be assigned to 2 groups and administered a lower single dose tablet (Period 1). After one week's wash-over period, the volunteers take higher dosages (Period 2).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males subjects, 20-45 years inclusive
* Weight over 55 kg inclusive and Ideal Body Weight (IBW) between -20% and +20% inclusive
* Written informed consent given

Exclusion Criteria:

* Hypersensitivity to drugs(aspirin, antibiotics and so on) including naftopidil
* History or presence of any clinically significant liver or kidney disease, gastrointestinal, cardiovascular, respiratory, endocrinal, musculoskeletal, neurologic/psychiatric, urinary, hematological, oncological pathology
* Have a history of drug abuse, or show positive for drug abuse at urine screening
* Have participated in another clinical study within 2 months prior to entering inth the study
* Are considered ineligible by the investigator due to clinical laboratory results or any other relevant reasons

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-09; Primary Completion 2009-10 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of naftopidil | Dec. 2009 (anticipated)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D.,Ph.D., Principal Investigator — Assistant Professor of Clinical Pharmacology, Seoul Nat'l Univ. Hospital
Locations (1):
- Clinical Trial center, Clinical Research institute, Seoul National University Hospital, Seoul, South Korea